CLINICAL TRIAL: NCT06747052
Title: Gender Impact on Physical Activity in Chronic Musculoskeletal Disorders Prevention: a Survey-based Cross-sectional Study in Regione Lombardia
Brief Title: Gender Impact on Physical Activity in Chronic Musculoskeletal Disorders Prevention
Acronym: Move4Health
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: WeMoveForHealth
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Musculoskeletal Disease; Gender Equity
Keywords: Physical activity; Gender; Musculoskeletal; Gender Equity; Surveys and Questionnaires; Cross-Sectional Studies
MeSH Terms: conditions — Motor Activity; Musculoskeletal Diseases; Coitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults residents in Lombardia Region: Adults with age ranging between 18 and 64 years, residents in Lombardia Region and spoken/reader Italian language

SUMMARY:
The goal of this survey based cross-sectional survey is to understand if there are gender patterns in physical activity participation and how they are associated with gendered organization of work and family activities, identifying socio-environmental variables that hamper the participation of both females and males in an active and healthy lifestyle. This survey also aim to explore if awareness and beliefs regarding musculoskeletal disorders and physical activity as factor for prevention differ according to gender and sex.

The main question is to investigate gender differences in physical activities participation in terms of adherence or not adherence to WHO recommendations by adjusting for socio-environmental variables.

The secondary questions are:

* To explore impact of gender on health status and sedentary behavior at same adherence and intensity level of physical activity
* To explore whether awareness and beliefs on musculoskeletal disorders and physical activity as prevention factor in the general population differ according to gender and sex.

DETAILED DESCRIPTION:
Musculoskeletal disorders rank high in global disease burden, with women disproportionately affected. Physical inactivity, a key modifiable risk factor for chronic diseases, is more prevalent among women globally, influenced by social and environmental factors. Despite initiatives like the WHO's Global Action Plan on Physical Activity, gender disparities persist, necessitating targeted interventions to enhance equitable physical activity participation and address associated healthcare costs, as exemplified by Italy's recent prevention efforts.

The aim of the current study is to understand if there are gender patterns in physical activity participation and how they are associated with gendered organization of work and family activities, identifying socio-environmental variables that hamper the participation of both females and males in an active and healthy lifestyle.

The survey will be developed using SurveyMonkey® software, an online survey management software. Following approval from the Ethics Committee, the survey will be shared to adults residing in the Lombardy Region (Italy) through direct contacts or online channels (e.g., emails, social networks, online via a dedicated project webpage) using an ad hoc generated link. Formal informed consent will be collected online before starting the survey. Participation in the survey will be anonymous and voluntary with no payoff. After recruitment, data will be collected using Microsoft Excel and stored at the IRCCS Ospedale Galeazzi - Sant'Ambrogio, Milan, Italy.

The theoretical framework will be built drawing on similar questionnaires published in the literature and leaded by international recognized organizations assessing public physical activity participation and knowledge and perceptions towards chronic musculoskeletal disorders. Three experts will pilot the prefinal draft of the survey to assess face and content validity on the prefinal draft of the survey. Experts' feedback will be used to introduce minor amendments to the survey.

The final questionnaire version consisted of five sections:

(i) Characteristics of the respondent and socio-environmental context (ii) Work life balance (iii) Lifestyle habits and physical activity (iv) Knowledge and perception of chronic MSK disorders and physical activity as a preventive factor.

(v) The SF-12 questionnaire to assess health status of the participants.

The sample size calculation will be based on assumptions on primary and secondary outcomes, considering the most conservative value as sample size of interest.

Specifically:

* Primary outcome: adherence to WHO recommendation Assuming an adherence to WHO recommendation (ie. Physical activity participation) among adult men of 40% and adult women of 30% (taken from ISTAT data of Lombardia Region), employing a 95% confidence, 80% power, the total sample size would be 712 adults. Only on this outcome we then considered different scenarios changing the expected percentage difference between men and women adherence to physical activity recommendation to 5% and 15%.
* Secondary outcome: difference in health status between women and men at the same level of physical activity Assuming a difference in heath status between women and men of 1,3 on SF12 (women SF12 = mean 44.5 ± 7.4, men SF12= mean 43.2 ± 7.8), a variability of 7.5, employing a 95% confidence, 80% power, the total sample size would be 1048 adults.
* Secondary outcome: difference in sedentary behavior between women and men at the same level of physical activity Assuming a difference in sedentary behavior between women and men of 0.94 hours per day (sedentary behavior man = 7.94 hours/day, sedentary behavior women = 8.89 hours/day), a variability of 2.13, employing a 95% confidence, 80% power, the total sample size would be 162 adults.

Overall, based on these calculations, 1048 adults will be needed as sample size that allow us to find a difference in adherence to physical activity of 10% between men and women but also guarantee a sufficient power for secondary outcomes.Taking into consideration non-responders and so an estimated response rate of 80% and a required sample size calculated in 1048 subjects, the number of individuals (out of the adult population residents in the Lombardy region of 6.371.890) needed to invite to participate at the survey to achieve the required sample size based on the expected response rate is 1310.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age range between 18 and 64 years, residents in Region Lombardia and spoken/reader Italian language

Exclusion Criteria:

* People with less than 18 years of age or more than 64 years of age. No other exclusion criteria will be applied.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents in Region Lombardia and spoken/reader Italian language
Sampling Method: Non-Probability Sample
Enrollment: 1310 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to WHO recommendations on physical activity | baseline (cross-sectional study)
  Gender differences in the prevalence of adherents to WHO recommendations on physical activity assessed as a dichotomous variable (adherent or non-adherent), based on responses to the questions: "Can you quantify the amount of time you spend doing regular physical activity per week?" and "Can you quantify the usual intensity level (moderate/vigorous) of your physical activity per week?"

SECONDARY OUTCOMES:
Health status | baseline (cross-sectional study)
  Gender differences in mean health status measured with the 12-item Short Form Survey (SF-12) questionnaire.
  The SF-12 is a multi-purpose, generic measure of health status that allows for the construction of summary measures that assess the physical (PCS) and mental (MCS) health status of the participant. Scores are calculated using an algorithm. A score of 50 or higher indicates good health, while a score below 50 suggests poor health.
Sedentary behavior | baseline (cross-sectional study)
  Gender differences in the prevalence of sedentary behavior assessed as a dichotomous variable (higher or lower than 6 sitting hours a day), based on responses to the question: "On a typical work or study day, how many hours do you spend sitting?"

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cule M, Guliani H. Are there gender based differences in participation and time spent in physical activity in Albania? Evidence from 2017-18 demographic and health survey. Arch Public Health. 2022 Aug 11;80(1):187. doi: 10.1186/s13690-022-00930-2. PMID 35953833
- [Background] Eizagirre-Sagastibeltza O, Fernandez-Lasa U, Yanci J, Romaratezabala E, Cayero R, Iturrioz I, Usabiaga O. Design and Validation of a Questionnaire to Assess the Leisure Time Physical Activity of Adult Women in Gipuzkoa. Int J Environ Res Public Health. 2022 May 8;19(9):5736. doi: 10.3390/ijerph19095736. PMID 35565129
- [Background] Oliveira AJ, Lopes CS, Rostila M, Werneck GL, Griep RH, Leon AC, Faerstein E. Gender differences in social support and leisure-time physical activity. Rev Saude Publica. 2014 Aug;48(4):602-12. doi: 10.1590/s0034-8910.2014048005183. PMID 25210819
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Ding D, Lawson KD, Kolbe-Alexander TL, Finkelstein EA, Katzmarzyk PT, van Mechelen W, Pratt M; Lancet Physical Activity Series 2 Executive Committee. The economic burden of physical inactivity: a global analysis of major non-communicable diseases. Lancet. 2016 Sep 24;388(10051):1311-24. doi: 10.1016/S0140-6736(16)30383-X. Epub 2016 Jul 28. PMID 27475266
- [Background] Liu S, Wang B, Fan S, Wang Y, Zhan Y, Ye D. Global burden of musculoskeletal disorders and attributable factors in 204 countries and territories: a secondary analysis of the Global Burden of Disease 2019 study. BMJ Open. 2022 Jun 29;12(6):e062183. doi: 10.1136/bmjopen-2022-062183. PMID 35768100
- See also: WHO Physical activity — https://www.who.int/news-room/fact-sheets/detail/physical-activity
- See also: WHO More active people for a healthier world The global action plan on physical activity 2018 - 2030 — https://www.who.int/initiatives/gappa
- See also: Piano regionale di prevenzione 2021 - 2025 Regione Lombardia — https://www.regione.lombardia.it/wps/portal/istituzionale/HP/DettaglioRedazionale/istituzione/direzioni-generali/direzione-generale-welfare/piano-regionale-prevenzione/piano-regionale-prevenzione
- See also: CDC Questionnaires, Datasets, and Related Documentation — https://archive.cdc.gov/#/details?url=https://www.cdc.gov/nchs/nhis/physical_activity/pa_questionnaires.htm